CLINICAL TRIAL: NCT06654336
Title: Phase II Randomized Trial of Recurrence-directed Therapy (RDT) With or Without Androgen-Deprivation Therapy (ADT) In Radio-recurrent Oligo-metastatic Hormone/Castrate Sensitive Prostate Cancer (romCSPC).
Brief Title: Study of Recurrence-directed Therapy (RDT) With or Without Androgen-Deprivation Therapy (ADT) In Patients With Radio-recurrent Oligo-metastatic Hormone/Castrate Sensitive Prostate Cancer (romCSPC)
Acronym: RATIONAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2024-RATΙONAL
Record Dates: First submitted 2024-10-16; First posted 2024-10-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma; Castration Sensitive Prostate Cancer
Keywords: Prostate adenocarcinoma; Castration Sensitive Prostate Cancer; Recurrent Oligo-metastatic Castration Sensitive Prostate CancerSPC; Andrigen Deprivation Therapy; Eligard; Recurrence Directed Therapy; Radiotherapy; Bio-chemical recurrence; Androgen Deprivation Therapy
MeSH Terms: interventions — luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recurrence-directed therapy (RDT) + ADT x 12 months (Experimental): Local, regional or distant oligometastatic RDT in addition to treatment with ADT for 12 months in the form of ELIGARD®.
  Interventions: Radiation: Recurrence-directed therapy (RDT); Drug: ELIGARD 22.5mg
- Recurrence-directed therapy (RDT) alone (Active Comparator): Local, regional, and distant oligometastatic RDT.
  Interventions: Radiation: Recurrence-directed therapy (RDT)

INTERVENTIONS:
Radiation: Recurrence-directed therapy (RDT) — RDT options include radiotherapy or surgical resection.
Drug: ELIGARD 22.5mg — ADT in the form of ELIGARD 22.5 mg every 3 months for a total of 12 months.
  Arms: Recurrence-directed therapy (RDT) + ADT x 12 months

SUMMARY:
The goal of this study is to determine whether the addition of Androgen Deprivation Therapy (ADT) utilizing the study drug ELIGARD® to Recurrence- Directed Therapy (RDT) improves progression-free survival (PFS) compared to RDT alone in patients with early radio-recurrent oligo-metastatic castrate / hormone sensitive prostate cancer (romCSPC). Participants will be assessed at standard of care clinic visits every 3 months. The follow-up period is 36 months.

DETAILED DESCRIPTION:
A multi-centre, open-label, phase II randomized clinical trial evaluating the addition of Androgen Deprivation Therapy (ADT) utilizing the study drug ELIGARD® compared to Recurrence Directed Therapy (RDT) alone in patients with previously localized prostate adenocarcinoma treated with definitive radiotherapy or with salvage radiotherapy after radical prostatectomy who experience biochemical recurrence and present with oligo-metastases (i.e., < 5 sites of metastases) on conventional imaging. Eligible and consenting patents will be randomized in a 1:1 fashion to either RDT alone (standard arm) or RDT +ADT (ELIGARD®) x12 months (experimental arm). During treatment study participants will be assessed for disease progression, development of castrate resistant prostate cancer (CRPC), acute and late genitourinary (GU) and gastrointestinal (GI) radiotherapy toxicity, the occurrence of adverse events, initiation of tertiary therapy, overall survival and quality of life through the completion of participant questionnaires. Participants will be assessed at standard of care clinic visits every 3 months. The follow-up period is 36 months from the date of randomization. The planned sample size is 162 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Previous biopsy-proven localized prostate adenocarcinoma (without predominant features of sarcomatoid, small cell or neuroendocrine carcinoma) treated with definitive or salvage radiotherapy ≥ 2 years or more before enrollment.
2. Recurrent Oligo-metastatic CSPC, M0 on conventional imaging (bone scan and CT scan of chest/abdomen/pelvis) with ≤ 5 metastases cumulative on all imaging, including MRI and PSMA-PET.

   Note: Patients with conventional imaging M1 oligometastatic CSPC, who have no more than 5 metastatic sites in all imaging modalities including MRI and PSMA-PET, will be accepted for study enrollment.
3. All sites of recurrent disease must be amenable to treatment with radiotherapy or surgery in the judgment of the investigator.
4. Biochemical recurrent prostate cancer with ONE of the following PSA recurrence definitions:

   1. After definitive radiotherapy (prostate in situ), with PSA ≥ nadir + 2ng/ml;
   2. After prostatectomy and adjuvant/salvage radiotherapy, with PSA ≥ nadir + 0.2ng/ml.

Exclusion Criteria:

1. Age < 18.
2. ECOG Performance Status ≥3.
3. PSA ≥ 20 ng/ml.
4. Treatment with ADT within 2 years from study enrollment or treatment with any androgen receptor axis within 6 months from study enrollment.
5. Prior treatment with chemotherapy for prostate cancer or bilateral orchiectomy. Note: prior chemotherapy for a different type of cancer is allowed if the patient has been continuously disease-free for > 3 years.
6. Intracranial or intrathecal metastasis.
7. Spinal cord compression, or spinal intramedullary metastasis.
8. Prior malignancy (except non metastatic, non- melanomatous skin cancer) unless disease free for > 3 years.
9. Bilateral hip prosthesis, treated earlier with definitive prostate radiotherapy, who have evidence of local disease recurrence within the prostate and no option for salvage treatment with brachytherapy or surgery.
10. Previous documented hypersensitivity to ELIGARD® or other GnRH agonist analogs of components of such preparations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Composite progression free survival | Time from randomization to the occurrence of composite PFS event occurring up to the 36 month follow-up.
  Biochemical, radiological or clinical progression [composite PFS (cPFS) event]

SECONDARY OUTCOMES:
Disease progression | Time from date of randomization, until the date of progression or death occurring up to the 36 month follow-up.
  Disease progression: time to biochemical progression (bPFS) (proportion of bPFS events); Disease progression: proportion of conventional-imaging based progression (rPFS) (proportion of rPFS events); Disease progression: proportion with eugonadal progression (egPFS)
Time to initiation of tertiary therapy; | Time of initial therapy to 36 month follow-up.
  Any non-protocol treatment given for prostate cancer after protocol-specified intervention.
Proportion of patients that develop castrate-resistant prostate cancer (CRPC) | During the 36 month follow-up.
  Proportion of patients that develop castrate-resistant prostate cancer (CRPC)
Overall survival. | During the 36 month follow-up.
  Overall survival.
Rate of early and late Grade 3 or higher GU and GI toxicity. | At 3, 6, 15 and 36 months.
  The rate of early and late Grade 3 or higher GU and GI toxicity will be assessed at baseline, 3, 6, 15 and 36 months. The CTCAEv.5.0 (> Grade 3, GI and GU) toxicity rates will be reported.
Quality of life assessed by EORTC QLQ C30 | Completed by the study participant at scheduled follow-up visits (Months 3, 6, 15 and 36).
  Study participant reported quality of life utilizing the following measurement EORTC QLQ C30
Quality of life assessed by EORTC QLQ PR25 questionnaire | Completed by the study participant at scheduled follow-up visits (Months 3, 6, 15 and 36).
Quality of life assessed by EORTC QLQ PRT20 questionnaire | Completed by the study participant at scheduled follow-up visits (Months 3, 6, 15 and 36).

CONTACTS AND LOCATIONS:
Overall Officials: Theos Tsakiridis, Dr., Principal Investigator — McMaster University; Jim Wright, Dr., Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes
A complete de-identified patient-level data set will be made available to academic affiliated researchers for the purpose of meta-analysis or a newly proposed study.
  * Data will be made available following submission of a maximum 2-page proposal. The study Steering Committee will review and, if acceptable, provide approval of the request.
  * A signed data sharing access/transfer agreement will be required between the requesting party and OCOG.
  * Authorship of publications to include the name of the study Principal Investigator.
  * The data will be provided as SAS datasets (as a CPT or XPT file). Any other format requests or additional statistical support may incur costs to the requestor.
  * Data will become available 12 months after publication by the study Principal Investigator, of the initial study results
Supporting Information: Analytic Code
Time Frame: Data will become available 12 months after publication by the study Principal Investigator, of the initial study results.
  Note: The timeframe may vary based on the journal and internal contractual obligations. The relevant timeframe should be adjusted accordingly to be study specific.
Access Criteria: A complete de-identified patient-level data set will be made available to academic affiliated researchers for the purpose of meta-analysis or a newly proposed study.
  * Data will be made available following submission of a maximum 2-page proposal. The study Steering Committee will review and, if acceptable, provide approval of the request.
  * A signed data sharing access/transfer agreement will be required between the requesting party and OCOG.
  * Data requests should be submitted to the OCOG Director.
URL: https://www.ocog.ca/PORTAL/Site/Home